CLINICAL TRIAL: NCT06901219
Title: The Effect of Fatigue on Static and Dynamic Balance in Healthy Young Male Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuwait University (Other)
Responsible Party: Principal Investigator, Dr. Anwar Amutairi, Assistant Professor, Kuwait University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: no. BE-17-14
Record Dates: First submitted 2025-03-16; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Fatigue
Keywords: Static Balance; Athletes; Dynamic Balance; Lactate
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fatigue protocol group (Experimental): The experimental group went through a fatigue protocol, in which speed and incline increase one unit each minute passing, and stopped when rate of perceived exertion level reached ≥ 18, and the plasma lactate level differed from the baseline by ≥ 4mmol/L
  Interventions: Behavioral: Running Fatigue Protocol
- Control (No Intervention): Will rest for 20 minutes

INTERVENTIONS:
Behavioral: Running Fatigue Protocol — The experimental group went through a fatigue protocol, in which speed and incline increase one unit each minute passing, and stopped when rate of perceived exertion level reached ≥ 18, and the plasma lactate level differed from the baseline by ≥ 4mmol/L.
  Arms: Fatigue protocol group

SUMMARY:
Participants were randomized into control and experimental groups. They were examined on static and dynamic balance (pre- & post-tests). Then, the experimental group went through a fatigue protocol, in which speed and incline increase one unit each minute passing, and stopped when rate of perceived exertion level reached ≥ 18, and the plasma lactate level differed from the baseline by ≥ 4mmol/L.

ELIGIBILITY:
Inclusion Criteria:

* male and aged between 18-24 years old,
* physically active (i.e. exercised ≥ 3 times weekly during the past three months).

Exclusion Criteria:

* reported a minor injury in the past two months,
* major injury in the past 12 months, and/or underwent a major primary surgery in their lower limb.

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Dynamic Balance | Baseline and immediately after the protocol
  Dynamic postural balance was measured using Y-balance (YB). A test designed to examine the ability to maintain postural stability in dynamic conditions. In this test, participants would single-leg stand on a block (start with left) and were instructed to push another block with their other leg as far as they can without losing their balance (i.e. placing their leg on the ground), while having their hands on their hips. The free blocks are placed anteriorly and posterolaterally of the participant in both directions, creating a Y shape with the stable block on the intersection of these lines. Distance reached was recorded for each direction. The directions of the test were anterior, posteromedial, posterolateral (pushing on the contralateral side). Then, the participants were asked to switch their feet and preform the task again; six trials in total were recorded to minimize learning effect.
Static balance | Baseline and immediately after the protocol
  Static balance (SB) testing was performed using virtual reality interactive gaming system (Wii balance board (WBB) [Nintendo, Kyoto, Japan]). The WBB contains four strain gauge-based load sensors, qualified to obtain center of pressure movement, which makes it valid and reliable to measure posture stability5. The participants were asked to perform stand quietly with their hand on their sides with both legs with equal weight-bearing and on a single-leg stance on the right leg, then on the left leg. All postures were performed under two conditions: open eyes and closed eyes.

CONTACTS AND LOCATIONS:
Locations (1):
- Kuwait University, Safat, Kuwait

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wikstrom EA. Validity and reliability of Nintendo Wii Fit balance scores. J Athl Train. 2012 May-Jun;47(3):306-13. doi: 10.4085/1062-6050-47.3.16. PMID 22892412
- [Background] Clark RA, Mentiplay BF, Pua YH, Bower KJ. Reliability and validity of the Wii Balance Board for assessment of standing balance: A systematic review. Gait Posture. 2018 Mar;61:40-54. doi: 10.1016/j.gaitpost.2017.12.022. Epub 2017 Dec 30. PMID 29304510
- [Background] Kluger BM, Krupp LB, Enoka RM. Fatigue and fatigability in neurologic illnesses: proposal for a unified taxonomy. Neurology. 2013 Jan 22;80(4):409-16. doi: 10.1212/WNL.0b013e31827f07be. PMID 23339207
- [Background] Bogdanis GC. Effects of physical activity and inactivity on muscle fatigue. Front Physiol. 2012 May 18;3:142. doi: 10.3389/fphys.2012.00142. eCollection 2012. PMID 22629249
- [Derived] Almutairi AB, Alabdulwahab A, Alkhalidi M, Alnouri S, Alkatan M. The effect of fatigue on static and dynamic balance in healthy young male athletes: a randomized trial. BMC Sports Sci Med Rehabil. 2025 Oct 31;17(1):316. doi: 10.1186/s13102-025-01363-4. PMID 41174785